CLINICAL TRIAL: NCT07060638
Title: Integrated Therapies for Alcohol Use in Alcohol-associated Liver Disease (ITAALD) Trial
Acronym: ITAALD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samer Gawrieh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Samer Gawrieh, Professor of Medicine. Director, Hepatology Clinical and Research Fellowship Program Clinical Director, NIAAA Alcoholic Hepatitis Network DCC, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITAALD; U24AA026969 (NIH)
Record Dates: First submitted 2025-06-10; First posted 2025-07-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Alcohol-associated Hepatitis
Keywords: Severe AH, AUD
MeSH Terms: interventions — Interleukin-22; eflepedocokin alfa; Prednisone; Acamprosate; Motivational Interviewing; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IL-22 (F-652), Prednisone Placebo, Acamprosate, MI and MET (Active Comparator): F-652 on days 1 and 7 and matching placebos for prednisone for 28 days and acamprosate for 6 months. MI will be delivered during the hospitalization; MET sessions will be delivered in the first 3 months
  Interventions: Drug: IL-22; Drug: Acamprosate; Drug: Prednisone placebo; Behavioral: Motivational Interviewing (MI); Behavioral: Motivational Enhancement Therapy (MET)
- IL-22 (F-652), Prednisone Placebo, and usual care (Active Comparator): F-652 on days 1 and 7 and matching placebo for prednisone for 28 days and usual care for AUD.
  Interventions: Drug: IL-22; Drug: Prednisone placebo; Behavioral: Usual Care
- Prednisone, IL-22 (F-652) Placebo, Acamprosate, MI, and MET (Active Comparator): Prednisone for 28 days and matching placebos for F-652 on days 1 and 7 and acamprosate for 6 months. MI will be delivered during the hospitalization; MET sessions will be delivered in the first 3 months
  Interventions: Drug: Prednisone; Drug: Acamprosate; Drug: IL-22 (F-652) Placebo; Behavioral: Motivational Interviewing (MI); Behavioral: Motivational Enhancement Therapy (MET)
- Prednisone, IL-22 (F-652) Placebo, and usual care (Active Comparator): Prednisone for 28 days and matching placebo for F-652 on days 1 and 7 and usual care for AUD.
  Interventions: Drug: Prednisone; Drug: IL-22 (F-652) Placebo; Behavioral: Usual Care

INTERVENTIONS:
Drug: IL-22 — F-652 (IL-22) is a fusion protein of human IL-22 with IgG2 fragment, and has anti-inflammatory effects
  Other Names: F-652
  Arms: IL-22 (F-652), Prednisone Placebo, Acamprosate, MI and MET; IL-22 (F-652), Prednisone Placebo, and usual care
Drug: Prednisone — Prednisone is an adrenal glucocorticoid with anti-inflammatory effects
  Arms: Prednisone, IL-22 (F-652) Placebo, Acamprosate, MI, and MET; Prednisone, IL-22 (F-652) Placebo, and usual care
Drug: Acamprosate — Acamprosate is a propane-1 sulfonic acid with anti-ethanol dependency effects
  Arms: IL-22 (F-652), Prednisone Placebo, Acamprosate, MI and MET; Prednisone, IL-22 (F-652) Placebo, Acamprosate, MI, and MET
Drug: Prednisone placebo — Matching placebo
  Other Names: Placebo
  Arms: IL-22 (F-652), Prednisone Placebo, Acamprosate, MI and MET; IL-22 (F-652), Prednisone Placebo, and usual care
Drug: IL-22 (F-652) Placebo — Matching Placebo
  Other Names: Placebo
  Arms: Prednisone, IL-22 (F-652) Placebo, Acamprosate, MI, and MET; Prednisone, IL-22 (F-652) Placebo, and usual care
Behavioral: Motivational Interviewing (MI) — MI is an evidence-based counseling style to overcome ambivalence to treatment in AUD patients
  Other Names: Behavioral therapy
  Arms: IL-22 (F-652), Prednisone Placebo, Acamprosate, MI and MET; Prednisone, IL-22 (F-652) Placebo, Acamprosate, MI, and MET
Behavioral: Motivational Enhancement Therapy (MET) — MET is an MI-based approach that includes 2-4 behavioral treatment sessions based on the Platform Treatment Manual
  Other Names: Behavioral therapy
  Arms: IL-22 (F-652), Prednisone Placebo, Acamprosate, MI and MET; Prednisone, IL-22 (F-652) Placebo, Acamprosate, MI, and MET
Behavioral: Usual Care — defined as a brief intervention with advice not to drink alcohol-containing beverages and referral to a 12-step program
  Arms: IL-22 (F-652), Prednisone Placebo, and usual care; Prednisone, IL-22 (F-652) Placebo, and usual care

SUMMARY:
This is a multicenter, randomized, double-blinded, placebo-controlled trial focused on the treatment of severe alcohol-associated hepatitis (sAH) and alcohol use disorder (AUD).

The primary purpose of the study is to determine whether subjects receiving sAH therapy in addition to AUD treatments will have better alcohol and liver-related outcomes at 6 months compared to sAH therapy plus usual care for AUD. Patients assigned to the AUD treatment will receive Acamprosate and counseling whereas those assigned to AUD standard care will receive brief advice and referral to a 12-step program.

The secondary purpose of the study is to determine if F-652 is safe and effective in treating sAH when compared to prednisone. Subjects will receive F-652 on days 1 and 7 or prednisone for 28 days. Outcomes will be measured by overall survival at 90 days.

DETAILED DESCRIPTION:
Objectives:

1. To determine whether interventions directed to treat AUD integrated with sAH therapies will improve a composite endpoint of alcohol and liver-related events at 6 months compared to usual care for AUD (primary endpoint).
2. To compare 90-day survival in patients receiving F-652 with those receiving up to 28 days of prednisone using the Day-7 Lille score as a stopping rule (secondary endpoint).
3. To compare one-year overall survival in patients receiving either IL-22 or prednisone with or without acamprosate (secondary endpoint).

Trial design and conduct

The Investigators will conduct a prospective, multicenter, sequentially randomized trial in 216 patients with sAH using a sequentially randomized design for proof of concept. The trial will assess whether integrated treatment of sAH and AUD reduces alcohol- and liver-related events and mortality.

The trial design resembles a 2X2 factorial study, but the AUD treatment assignment [acamprosate + motivational interviewing (MI) + motivational enhancement therapy (MET)] versus usual care (UC), defined as a brief intervention with advice not to drink alcohol-containing beverages and referral to a 12-step program, is done on Day 7 after the start of the sAH treatment. Only survivors of the first 7 days will be randomized to receive the AUD intervention or UC.

The study will be conducted at six clinical sites in the United States selected by the National Institute of Alcoholic Abuse and Alcoholism (NIAAA) and supported by a Data Coordinating Center at Indiana University (DCC). The DCC will also manage the biorepository.

The study will be conducted according to Good Clinical Practice (GCP) and in compliance with local, state, and federal regulatory requirements. Adverse events during the trial will be identified, recorded, assessed for causality, and reported in accordance with FDA guidance. In addition to general assessment, the investigators will specifically focus on (1) rates and types of infection as well as their severity, (2) potential development of drug-induced liver injury, (3) injection site reactions, and (4) hematological adverse events.

This study will be approved by an appropriately convened single IRB, Advarra, and will be monitored by an NIAAA-appointed Data and Safety Monitoring Board (DSMB). The Investigators will conduct this study under an Investigational New Drug (IND) application from the United States Food and Drug Administration (FDA).

It is anticipated that a centrally located investigational pharmacy at Indiana University will dispense the study medications to all participating sites under close coordination from the DCC. The study will provide the participants with F-652, prednisone, matching placebos, and acamprosate.

Duration of Trial by Phase Treatment phase: up to 6 months Follow-up phase: up to two years

Interventions to be tested F-652 vs. prednisone as treatment for sAH. AUD interventions (acamprosate + MI + MET) versus usual care for AUD treatment.

Group assignment:

The Investigators will sequentially randomize the study participants into four treatment groups.

On day 1, participants will be randomized to receive either F-652 or prednisone at a 1-to-1 ratio. Those randomized to receive F-652 will also receive a prednisone placebo; those randomized to receive prednisone will receive the F-652 placebo. Prednisone or prednisone placebo will be stopped if the Day-7 Lille score is >0.45.

On day 7, survivors will be randomized to receive either the AUD intervention (acamprosate + MI + MET) or usual care at a 1-to-1 ratio.

Block randomization will be used to ensure balanced group sizes in randomization.

So, there will be four treatment combinations:

ARM 1: F-652 on days 1 and 7 and matching placebos for prednisone for 28 days and acamprosate for 6 months. MI will be delivered during the hospitalization; MET sessions will be delivered in the first 3 months.

ARM 2: F-652 on days 1 and 7 and matching placebo for prednisone for 28 days and usual care for AUD.

ARM 3: Prednisone for 28 days and matching placebos for F-652 on days 1 and 7 and acamprosate for 6 months. MI will be delivered during the hospitalization; MET sessions will be delivered in the first 3 months.

ARM 4: Prednisone for 28 days and matching placebo for F-652 on days 1 and 7 and usual care for AUD.

Distribution of study drug and placebo Participants or guardians will be instructed on drug timing and dose of these experimental treatments after discharge from the hospital. Study personnel will ensure participants and guardians are knowledgeable about the frequency and amount before the end of the study visit, and an instructional document will be provided.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18, <70
* MELD 20-35 on day of randomization
* Definitive or probable diagnosis as defined by the NIAAA criteria
* Onset of jaundice (defined as serum total bilirubin >3 mg/dL) within the prior 8 weeks
* Ongoing consumption of > 40 gm (for females) and > 60 gm (for males) alcohol daily for 6 months or more with less than 8 weeks of abstinence before onset of jaundice
* AST > 50 IU/L,
* AST: ALT > 1.5
* ALT and AST values < 400 IU/L
* and/or histological evidence of AH*

  *In patients with possible AH or AH with confounding factors such as possible ischemic hepatitis, possible DILI, uncertain history of alcohol use (e.g., patient denies excessive alcohol use), and atypical/abnormal laboratory tests (e.g., AST < 50 IU/L or > 400 IU/L, AST/ALT ratio < 1.5), antinuclear antibody > 1:160 or SMA > 1:80, a standard of care liver biopsy may be performed during current hospital admission to confirm AH and exclude competing etiologies.
* Females of childbearing (reproductive) potential must have a negative serum or urine pregnancy test at screening.

Exclusion Criteria

* Active listing for liver transplantation before screening
* MELD score <20 or > 35
* Uncontrolled infection (persistent positive blood or other body fluid cultures despite 48 hours of antibiotic therapy)
* Progressive hemodynamic compromise requiring intravenous pressors
* Pneumonia as evidenced by clinical and radiological examination
* Renal failure defined by estimated GFR <35 mL/min.
* Clinically active C. diff infection
* Evidence of other liver diseases (such as autoimmune hepatitis, primary biliary cholangiopathy, primary sclerosing cholangitis, ischemic, sepsis- or drug-induced liver disease)
* History or presence of cancer (including hepatocellular carcinoma) other than non- melanoma skin cancer
* Prior exposure to systemic corticosteroid (glucocorticoid) or immunosuppressive therapy for more than 2 days within the previous 30 days
* Current use of naltrexone or acamprosate.
* Clinically significant pancreatitis- abdominal pain, elevated lipase (> 3 X ULN), and at least edema of pancreas with fat-stranding on CT scan
* Active gastrointestinal bleeding defined as hematemesis or melena with a decrease in hemoglobin more than 2 g/dl in 24 hours due to gastrointestinal bleeding, or with a decrease in mean arterial BP to < 65 mmHg
* Significant concomitant medical illnesses (such as uncontrolled congestive heart failure or COPD or progressive multi-organ failure) as determined by the study investigator
* Uncontrolled mental illness as determined by the study investigator
* Uncontrolled HBV, HIV, or HCV infection with persistent viremia. However, subjects with controlled (undetectable viral load) HIV and HBV on viral suppressive therapies will be enrolled and subjects with history of HCV will be enrolled if they have evidence of SVR one year prior to enrollment
* Active illicit opiates, cocaine, ketamine, or methamphetamine use in the last 30 days.
* Uncontrolled diabetes mellitus with A1c > 9
* Pregnancy or breastfeeding
* Known allergy or intolerance to therapeutic agents to be tested
* Unwillingness to stop alcohol use and to undergo AUD treatment
* Unwillingness to either abstain from sexual intercourse, or if sexually active, use a reliable method of birth control during the study and for at least 30 days after the last dose of the study medication. Examples of acceptable birth control methods include double barrier method such as condom and occlusive cap (diaphragm or cervical cap) with spermicidal foam/gel/film/cream/suppository; birth control pills, patches, injections, or implants; intrauterine device (IUD); vasectomy and tubal ligation.
* Participant has any condition or circumstance that adversely affects the participant, could cause noncompliance with treatment or visits, may impact the interpretation of clinical data, could cause bias, or may otherwise contraindicate the participant's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Death | 6 months
  Number (%) of participants who die from any cause
Liver transplant | 6 months
  Number (%) of participants who receive liver transplant
Ascites | 6 months
  Number (%) of participants with new onset of clinically detectable
Hepatic encephalopathy | 6 months
  Number (%) of participants with hepatic encephalopathy ≥ New Haven grade 2
Portal hypertensive bleeding | 6 months
  Number (%) of participants with gastroesophageal varices or portal gastropathy
Liver-related hospital admission | 6 months
  Number (%) of participants with liver-related hospital admission for ascites, hepatic encephalopathy, infection, GI bleeding
Increase in MELD score > 5 points | 6 months
  Number (%) of participants with increase in MELD score > 5 points
Return to drinking | 6 months
  Number (%) of participants that return to drinking defined as <100% abstinence-using timeline follow back questionnaire

SECONDARY OUTCOMES:
Transplant-free survival | 30 days, 90 days, 180 days, 1 year, and 2 years
  Time participants live without liver transplant

OTHER OUTCOMES:
Change in MELD Score | 30, 90, 180 days
  Increase or decrease in MELD score. MELD is Model for End-stage Liver Disease Model. Higher MELD is associated with worse outcomes while lower MELD is associated with better outcomes. MELD typically ranges from 6-40.
Acute kidney injury (AKI) | 30, 90, 180 days
  Number (%) of participants with AKI
Multi-organ failure | 30, 90, 180 days
  Number (%) of participants with multi-organ failure
Transfer to ICU | 30, 90, 180 days
  Number (%) of participants with transfer to ICU
Infection and sepsis | 30, 90, 180 days
  Number (%) of participants with infection and sepsis

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia